CLINICAL TRIAL: NCT05431803
Title: Real-World Study of Lanreotide Autogel for the Treatment of Patients With Acromegaly in China
Brief Title: Real-World Study (RWS) of Lanreotide Autogel (LAN) for the Treatment of Patients With Acromegaly in China
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52030-455
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the one-year effectiveness and safety of LAN among patients with acromegaly in China in routine clinical practice. In addition, the study is designed to understand the real-world treatment patterns and outcomes of LAN among Chinese patients with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are able to comply with the protocol
* Participants with serum IGF-1 level above the ULN for age and sex, and serum fasting GH level above 2.5 μg/L
* Participants with acromegaly who are naïve to LAN treatment and about to initiate LAN

Exclusion Criteria:

* Participants who are currently participating in any investigational study or clinical trial of acromegaly
* Pregnant participants
* Participants with hypersensitivity to somatostatin or related peptides or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants who have been diagnosed with acromegaly and initiating LAN treatment
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving full biochemical control | At 12 months
  Defined as fasting Growth Hormone (GH) ≤ 2.5 μg/L and Insulin-like Growth Factor-1 (IGF-1) normalization

SECONDARY OUTCOMES:
Percentage of participants achieving fasting GH < 1 μg/L and IGF-1 normalization | At 12 months
Percentage of participants achieving fasting GH ≤2.5 μg/L and IGF-1 ≤1.3 Upper Limit of Normal (ULN) | At 12 months
Mean change in fasting GH and IGF-1 concentrations. | From baseline to 3, 6, and 12 months
Mean change in the proportion of patients experiencing each of the symptoms (headache, excessive sweating, joint pain, fatigue, and soft tissue swelling) as evaluated by physicians. | From baseline to 6 and 12 months
Mean change in Quality of Life (QoL) scores | From baseline to 6 and 12 months
  Assessed by the Acromegaly Quality of Life Questionnaire (AcroQoL).
Treatment utilisation of LAN, evaluated by the total number of injections received | From baseline to 12 months
Treatment utilisation of LAN, evaluated by number of participants in Extended Dosing Interval (EDI) | From baseline to 12 months
Incidence of all Adverse Events (AEs) | From baseline to 3, 6 and 12 months
  Including Serious Adverse Events (SAEs) and special situations assessed according to incidence, intensity, causality, outcome, action taken, and seriousness.
Mean change in physical examination results | From baseline to 3, 6, and 12 months
  Including Body Mass Index (BMI) and weight
Mean change in vital signs blood pressure | From baseline to 3, 6, and 12 months
Mean change in vital signs heart rate | From baseline to 3, 6, and 12 months
Mean change in Clinical laboratory assessments | From baseline to 6, and 12 months
  Including fasting blood glucose, glycated hemoglobin A1C (HbA1c), total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL, and triglycerides
Mean change in free thyroxine (FT4) and cortisol for males and females | From baseline to 6 and 12 months
Mean change in testosterone for males only | From baseline to 6 and 12 months
Mean change in follicle-stimulating hormone (FSH), luteinizing hormone (LH), and estradiol for females only. | From baseline to 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (12):
- China (12):
  - Peking Union Medical College Hospital (PUMCH), Beijing
  - Peking University Third Hospital (PUH3), Beijing
  - Xiangya Hospital Central South University (XYHCSU), Changsha
  - West China Hospital，Sichuan University (WCH), Chengdu
  - The First Affiliated Hospital,Sun Yat-sen University (FAHSYSU), Guangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine (SAHZU), Hangzhou
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School (NJDTH), Nanjing
  - The First Hospital of China Medical University (CMU1H), Shenyang
  - The Second Hospital of Hebei Medical University (HB2H), Shijiazhuang
  - Affiliated Hospital of Wenzhou Medical University (FAHWMU), Wenzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology (TJH HUST), Wuhan
  - The First Affiliated Hospital of Zhengzhou University (FAHZZU), Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/